CLINICAL TRIAL: NCT04029844
Title: A Prospective, Single Arm Clinical Investigation Evaluating Safety and Performance of the Colibri Transcatheter Aortic Heart Valve System for the Treatment of Symptomatic Severe Aortic Stenosis Via Transfemoral Access in High Surgical Risk Patients
Brief Title: Colibri Transcatheter Aortic Heart Valve System Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colibri Heart Valve LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: COL-01
Record Dates: First submitted 2019-07-19; First posted 2019-07-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Severe Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Colibri Device (Experimental): Treatment
  Interventions: Device: Colibri TAVI System

INTERVENTIONS:
Device: Colibri TAVI System — Implantation of Colibri heart valve

SUMMARY:
The Colibri Heart Valve clinical investigation ("COL-01") is a prospective, multicenter, exploratory single arm and controlled clinical investigation compared to recent historical results. This study will be conducted in about 7 European sites. The study will evaluate the safety and performance of the Colibri Transcatheter Aortic Heart Valve System for the treatment of symptomatic severe aortic stenosis via transfemoral access in high surgical risk patients.

30 subjects suffering from symptomatic severe aortic tricuspid valve stenosis and who are at high surgical risk (logistic EuroSCORE I > 20% or other risk factors not included in this score such as frailty, porcelain aorta, sequelae of chest radiation or logistic EuroSCORE I < 20% but considered at high risk by local Heart Team evaluation) will be enrolled in this clinical investigation.

The primary objective of this clinical investigation is to evaluate the all-cause mortality at 30 days post implantation. The secondary objectives are to evaluate the safety and performance of the investigational device at 30 days, 6 and 12 months, and 2, 3, 4, 5 years post implantation.

ELIGIBILITY:
Inclusion Criteria:

* 1. Subject of age > 75 years
* 2. Subject suffering from severe aortic tricuspid valve stenosis defined as follows: High-gradient aortic stenosis (mean pressure gradient across aortic valve > 40 mmHg or peak velocity > 4.0 m/s)
* 3. Subject has symptomatic aortic valve stenosis with New York Heart Association (NYHA) > Class II
* 4. Subject with a documented local Heart Team (HT) agreement of high surgical risk as described in the population
* 5. ECG-gated Multi-Slice Computed Tomographic (MSCT) measurements determined an aortic annulus > 22 mm and < 27.4 mm
* 6. Subject deemed eligible by a TAVI Centralized Case Review Committee (CRC)
* 7. Subject can understand the purpose of the clinical investigation, has signed voluntarily the informed consent form and is agreeing to the scheduled follow-up requirements

Exclusion Criteria:

* 1. Arterial aorto-iliac-femoral axis unsuitable for transfemoral access as assessed by conventional angiography and/or multidetector computed tomographic angiography (access vessel diameter incompatible with a 16F sheath introducer)
* 2. Aortic root anatomy condition or lesion preventing implantation or access to the aortic valve
* 3. Non-calcific acquired aortic stenosis
* 4. Native unicuspid/bicuspid aortic valve or congenital aortic valve abnormality
* 5. Previous implantation of heart valve in any position
* 6. Severe aortic regurgitation (> 3+)
* 7. Severe mitral regurgitation (> 3+)
* 8. Severe tricuspid regurgitation (> 3+)
* 9. Severe left ventricular dysfunction (Left Ventricular Ejection Fraction (LVEF) < 30%)
* 10. Echocardiographic evidence of intracardiac mass, thrombus or vegetation
* 11. Multi-vessel coronary artery disease (CAD) with a Syntax Score or residual Syntax Score > 22 and/or unprotected left main coronary artery
* 12. Cardiogenic shock
* 13. Untreated cardiac conduction disease in need of pacemaker implantation
* 14. Uncontrolled atrial fibrillation (resting heart rate (HR) > 120bpm)
* 15. Active and/or suspicion of endocarditis or ongoing sepsis
* 16. Blood dyscrasias defined as: leukopenia (White Blood Cells (WBC) < 1,000/mm3), thrombocytopenia (Platelets (PLT) < 50,000/mm3), history of bleeding diathesis or coagulopathy, or hypercoagulable states
* 17. Evidence of acute myocardial infarction (MI) less than 30 days before signing informed consent
* 18. Any need for emergency surgery
* 19. Recent (< 6 months of signing informed consent) CerebroVascular Accident (CVA) or Transient Ischemic Attack (TIA)
* 20. Symptomatic carotid or vertebral artery disease or successful treatment of carotid stenosis < 30 days prior to signing informed consent
* 21. Any active bleeding that precludes anticoagulation
* 22. Liver failure (Child-C)
* 23. End-stage renal disease requiring chronic dialysis or creatinine clearance < 20cc/min
* 24. Pulmonary hypertension (systolic pressure >80mmHg)
* 25. Severe Chronic Obstructive Pulmonary Disease (COPD) demonstrated by a Forced Expiratory Volume (FEV1) < 750cc
* 26. Refusal of blood transfusion
* 27. A known hypersensitivity or contraindication to all anticoagulation/anti-platelet regimens (or inability to be anticoagulated for the index procedure), to cobalt chromium, to porcine and/or collagen, to glutaraldehyde or contrast media
* 28. Any medical, social or psychological condition that in the opinion of the investigator precludes the subject from giving appropriate consent or adherence to the required follow-up procedures
* 29. Currently participating in another drug or device trial (excluding observational registries) for which the primary endpoint has not been assessed
* 30. Estimated life expectancy of less than 12 months
* 31. For females, pregnancy or intention to become pregnant prior to completion of all follow-up procedures
* 32. Inability to comply with the clinical investigation requirements
* 33. Subject under judicial protection, tutorship or curatorship (for France only)

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2021-09-15 (Actual); Primary Completion 2023-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Rate of all-cause mortality at 30 days post implantation | 30 Days

CONTACTS AND LOCATIONS:
Overall Officials: Bernard Chevalier, MD, Principal Investigator — Hopital Prive Jacques Cartier
Locations (5):
- France (3):
  - Institut Coeur Poumon, CHRU, Lille
  - Hôpital Privé Jacques Cartier, Massy
  - Clinique Pasteur, Toulouse
- United Kingdom (2):
  - Brighton & Sussex University Hospital, Roayl Sussex County Hospital, Brighton, East Sussex
  - Barts Heart Centre / St Bartholomew's Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided